CLINICAL TRIAL: NCT01746680
Title: Phase IV STudy of Tacrobell in Active Rheumatoid Arthritis
Brief Title: Efficacy and Safety Study of Tacrobell to Treat Rheumatoid Arthritis
Acronym: TIARA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: m308RAP11M
Record Dates: First submitted 2012-12-04; First posted 2012-12-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; RA; tacrolimus; Disease Activity Score 28; EULAR
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus with Methotrexate (Experimental): Subjects have tacrolimus per oral once daily with methotrexate for 24weeks. Tacrolimus increased dosing regimen: 1mg for 0~4 weeks, 2mg for 4 weeks~8 weeks, 3mg for 8 weeks~24 weeks
  Interventions: Drug: Tacrolimus with Methotrexate

INTERVENTIONS:
Drug: Tacrolimus with Methotrexate — Tacrolimus 1 mg for 0~week4, 2mg for week4~week8, 3mg for week8~week24 with MTX ≤20mg/week
  Other Names: TacroBell® with MTX

SUMMARY:
The aims of this study are to assess the efficacy and safety of tacrolimus in patients with active rheumatoid arthritis(RA). EULAR(European League Against Rheumatism) response at week 24 compared to baseline will be evaluated to assess the efficacy of Tacrolimus.

DETAILED DESCRIPTION:
A Phase IV, Open labeled, Multi-Center Trial to Assess the Efficacy and Safety of Tacrolimus(Tacrobell®)in patients with active rheumatoid arthritis(RA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥20years
* Signed and dated informed consent document indicating that the patient
* Women of childbearing potential must have a negative serum or urine pregnancy test at the screening visit. Except in the case of surgically sterile or amenorrhea for one year.
* Female patients must agree to use adequate contraception measures during the period of therapy which should be continued for 4 weeks.
* have RA and meet all of the following criteria; RA occurring ≥ 3months and less than 15 years and diagnosed based on 1987 ACR classification criteria for rheumatoid arthritis; Active RA patients with MTX and among them who has insufficiency response to DMARDs as defined DAS28>3.2 in active RA patient. Insufficiency response is defined despite MTX therapy for > 12 weeks, RA activity≥ more than moderate and confirmable during 12 weeks, sequence of taking MTX >7.5mg/week for more than 6 weeks; ESR≥28mm/h or CRP≥1.0mg/dl; Tender Joint Counts must be more than 6 and Swollen Joint Counts must be more than 3

Exclusion Criteria:

* Inflammatory joint diseases, Systematic inflammatory disease
* Prosthesis and had an event of infected in it.
* Medical history of chronic infection, moderate infection or possibly to life threatening or signs and symptoms of serious infection.
* Patients have received treatment with a live vaccine from baseline within 8 weeks.
* HBsAg positive and hepatitis C virus positive patient.
* Patients have a history of malignancy. (But, carcinoma in situ of the uterine cervix or basal cell carcinoma have been treated is allowed within 5years)
* Patients have cardiovascular disease or associated disease which is not controlled.
* uncontrollable blood sugar(HbA1C ≥8%) or required insulin.
* Patients with a history of operation on index knee joint which could have influence on the result and need to have surgery as determined by investigator.
* At screening, patients have laboratory result as defined by ; white blood cell(WBC) < 3,500/mm3, Absolute Neutrophil Count(ANC) < 1,500/mm3, Hemoglobin < 8.5g/dl, Platelet count(PLT) < 100,000/mm3, Serum creatinine >1.5*upper limit of normal or 2mg/dl, Total bilirubin > 2*upper limit of normal, aspartate aminotransferase(AST) > 2*upper limit of normal, alanine aminotransferase(ALT) > 2*upper limit of normal, alkaline phosphatase(ALP) > 2*upper limit of normal
* Patients on any other clinical trial or experimental treatment in the past 8weeks
* An impossible one who participates in clinical trial by investigator's decision

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline European League Against Rheumatism(EULAR) response at 24weeks | baseline, 24weeks

SECONDARY OUTCOMES:
Change from baseline Simplified Disease Activity Index(SDAI) at 24weeks | baseline, 24weeks
Change from baseline Korean Health Assessment Questionnaire(KHAQ-20) at 24weeks | baseline, 24weeks
Change from baseline Erythrocyte Sedimentation Rate(ESR) at 16weeks | baseline, 16weeks
Change from baseline Erythrocyte Sedimentation Rate(ESR) at 24weeks | baseline, 24eeks
Change from baseline C-Reactive Protein(CRP) at 16weeks | baseline, 16weeks
Change from baseline C-Reactive Protein(CRP) at 24weeks | baseline, 24weeks
Change from baseline European League Against Rheumatism(EULAR) response at 16weeks | baseline, 16weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seung -Jae Hong, phD, Dr, Study Chair — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, South Korea